CLINICAL TRIAL: NCT05455242
Title: The Effectiveness of an Occupation-Based Habit Formation Intervention in Promoting Healthy Behaviors Among Individuals With Type 2 Diabetes
Brief Title: Habit Formation for Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Des Moines University (Other)
Responsible Party: Principal Investigator, Diana Feldhacker, Program Director and Department Chair, Des Moines University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-20-185
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Diabete Type 2
Keywords: Habit Formation; Occupational Therapy; Self-Management; Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Habit Formation Interventions (Experimental): Single subject design used for individual control (A-B design). During baseline phase (A), participants completed self-care activities ratings once per week for 4 weeks. During intervention phase (B), participants engaged in weekly sessions to address goals related to diabetes self-management and guided in habit formation. Participants engaged in intervention for 10 weeks, in accordance with habit formation recommendations by Lally et al. (2010). Each weekly session were held virtually (telephone or Zoom) and lasted 30-60 minutes, beginning with administration of the SDSCA and SRBAI. Participants were instructed in ongoing context-specific implementation intention to promote occupational participation in DSM through habit formation. This instruction included continued education and context modification recommendations. At two week intervals, additional areas of DSM were added until each were covered: blood glucose monitoring, nutrition, medication management, and physical activity.
  Interventions: Behavioral: Habit formation

INTERVENTIONS:
Behavioral: Habit formation — Habit formation interventions to promote context-dependent automatic behaviors to support diabetes self-management.

SUMMARY:
The purpose of the study is to determine the feasibility of interventions which focus on building habits as a method of improving diabetes self-management behaviors for individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old
* read and write in the English language
* have technology capability for virtual or telephone sessions
* are reachable by phone or text messaging
* have a diagnosis of T2DM
* were willing and able to participate in all study-related activities, and
* were not currently involved in other diabetes-related education and behavioral interventions.

Exclusion Criteria:

* younger than 19 years old
* unable to read and write in the English language
* did not have technology capability for virtual or telephone sessions
* were not reachable by phone or text messaging
* were unwilling or unable to participate in all study-related activities, and/or
* were currently receiving or involved in other diabetes-related education and behavioral interventions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Self-Care | 13 weeks
  The Summary of Diabetes Self-Care Activities (SDSCA) is a self-report questionnaire of DSM (diet, exercise, blood-glucose monitoring, foot care, and smoking) for which individuals report frequency of activities during the past 7 days (Toobert et al., 2000). A global self-care behavior score (average of items 1-10) was reported in days per week the participant executed self-care activities. In addition, combined subscales were used for general diet, specific diet, exercise, and blood glucose testing using a global average of items 1-8, reported in days per week. As part of baseline phase data collection (Phase A), the Summary of Diabetes Self-Care Activities (SDSCA) was administered once weekly for 4 weeks. Following the initial evaluation, interventions (phase B) were provided to participants once per week for 10 weeks and began with administration of the SDSCA.
Change in Behavior Automaticity | 10 weeks
  The Self-Report Behavior Automaticity Index SRBAI is a measure of habit strength and automaticity. Individuals respond how they perform a target behavior using a 7-point scale, with 7 meaning a better outcome. The initial evaluation session closed the baseline phase (Phase A) and initiated the intervention phase (Phase B) of the study. In this initial session, individuals were guided in setting a context-specific implementation intention for habit formation of a simple occupational habit related to nutrition. These nutrition intentions were utilized to create target behaviors for the Self-Report Behavioral Automaticity Index (SRBAI), which was administered at the end of the first session. Following the initial evaluation, interventions were provided to participants once per week for 10 weeks and began with administration of the SRBAI.

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No